CLINICAL TRIAL: NCT01353014
Title: Genetic Information and Dietary Intake Behaviour
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Advance Foods and Materials Network (Other)
Responsible Party: Principal Investigator, Ahmed El-Sohemy, Professor, University of Toronto
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: AElSohemy
Record Dates: First submitted 2011-05-04; First posted 2011-05-12 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
Keywords: Nutrigenomics; Diet; Nutrition
MeSH Terms: interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dietary advice with genetic information (Experimental): This group will receive dietary advice for caffeine, vitamin C, sugar and sodium based on genetic information.
  Interventions: Other: Dietary advice with genetic information
- General dietary recommendations (Active Comparator): This group will receive general dietary recommendations for caffeine, vitamin C, sugar and sodium from recognized health institutions (caffeine: Health Canada; sugar: the World Health Organization; vitamin C and sodium: the Institute of Medicine).
  Interventions: Other: General dietary recommendations

INTERVENTIONS:
Other: Dietary advice with genetic information — This group will receive dietary advice for caffeine, vitamin C, sugar and sodium based on genes that affect the metabolism of or sensitivity to caffeine, vitamin C, sugar and sodium.
  Arms: Dietary advice with genetic information
Other: General dietary recommendations — This group will receive general dietary recommendations from recognized health organizations for caffeine, vitamin C, sugar and sodium, with no genetic information.
  Arms: General dietary recommendations

SUMMARY:
This study's primary objective is to determine if providing individuals with personal genetic information impacts dietary intake behaviour. Specifically, the investigators will be examining whether providing dietary advice based on genes that affect the metabolism of or sensitivity to caffeine, vitamin C, sugar and sodium will impact the intake of these dietary components. The study hypothesis is that providing dietary advice based on genetics will impact dietary behaviour to a greater extent than general dietary recommendations.

ELIGIBILITY:
Inclusion Criteria:

* 20-35 year old participants from the Toronto Nutrigenomics and Health Study

Exclusion Criteria:

* pregnancy or nursing
* vitamin C supplement users
* caffeine intake < 100 mg/day
* total sugars intake < 10% energy
* sodium intake < 1500 mg/day

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 138 (Actual)
Dates: Start 2011-05; Primary Completion 2011-12 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Dietary Intake at 3 months | 3 months
  We will assess dietary intakes of caffeine (mg), vitamin C (mg), sugar (g and % energy) and sodium (mg) using Food Frequency Questionnaires (FFQ). An FFQ will be administered at baseline to determine dietary habits before dietary advice is given to either group (control or intervention). A second FFQ will be administered 3 months after the dietary advice is given, to examine if any changes were made to dietary intake in the short-term.
Change from Baseline in Dietary Intake at 12 months | 12 months
  A third FFQ will be administered 12 months after the dietary advice is given, to examine if any long-term dietary changes were made in intakes of caffeine (mg), vitamin C (mg), sugar (g and % energy) and sodium (mg).

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed El-Sohemy, PhD, Principal Investigator — University of Toronto
Locations (1):
- University of Toronto, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Nielsen DE, El-Sohemy A. Disclosure of genetic information and change in dietary intake: a randomized controlled trial. PLoS One. 2014 Nov 14;9(11):e112665. doi: 10.1371/journal.pone.0112665. eCollection 2014. PMID 25398084